CLINICAL TRIAL: NCT00292890
Title: Which Needle Length for Injecting Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1-Kreugel
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2005-01

CONDITIONS: Diabetes Mellitus
Keywords: injection devices; injection technique; insulin needles; insulin administration
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Device: insulin needle

SUMMARY:
Background and aims:

* In the Netherlands most patients with diabetes mellitus that are treated with insulin, use an insulin pen for insulin administration. The injection technique can influence the absorption rate of insulin.
* The aim of this study is to compare the effect of insulin injections using a 5 mm insulin needle with insulin injections using a longer needle, on HbA1c, bloodglucose levels, hypoglycaemic events, bleeding, bruising, insulin leakage and pain perception.
* Study Hypothesis: 'Insulin injected with needles of 5 mm can be given without a skinfold. The length of the needle will not influence HbA1c levels and bloodglucose levels'.

DETAILED DESCRIPTION:
* In this randomised, clinical trial with cross-over design, 52 patients with Diabetes type 1 and 2 using a 8 or 12 mm needle, are randomised into two groups.
* Group I starts using 5 mm needles for insulin administration, after 13 weeks group I returns to their previously used 8 or 12 mm needle
* Group II continues using their own 8 or 12 mm needle, after 13 weeks group II starts using 5 mm needles for insulin administration.
* During each visit the HbA1c level is measured and a copy is made of the logbook of the patient with the blood glucose measurements.
* Insulin doses and number of experienced hypoglycaemic events are registered at each visit.
* The opinion and experiences of the patients regarding the different needles are obtained by using a questionnaire.
* Within-group analyses are computed, using the Wilcoxon signed Ranks Test. Between-group analyses are computed using the Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* males and females diagnosed with diabetes Type 1 or 2
* using insulin for at least one year
* using an insulin pen and a needle of 8-mm or longer
* 18 years or older
* capable of reading the written information
* prepared to, and capable of signing an informed consent

Exclusion Criteria:

patients that

* change their own insulin dosage and don't keep an administration of these changes
* had an HbA1c that varied more than 15 % in the past year
* use a needle of 5 or 6-mm
* have hypoglycaemia unawareness
* are pregnant or wanted to become pregnant
* have a BMI < 18
* have a skinfold thickness of 10 mm or less at the injection sites (abdomen and thigh)
* had hemoglobinopathies which could limit the ability of haemoglobin to be glycated
* had skin problems like lipodystrofie

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-01; Study Completion 2004-10

PRIMARY OUTCOMES:
HbA1c levels, insulin doses and the number of experienced hypoglycaemic events

SECONDARY OUTCOMES:
blood glucose measurements and the experiences of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Bruce HR Wolffenbuttel, MD PhD, Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands